CLINICAL TRIAL: NCT02468323
Title: Prophylactic Antiemetic Efficacy of Palonosetron Versus Ondansetron for Cesarean Sections Under Regional Anesthesia: Study Single Center, Prospective, Double-blind, Randomized, Placebo Controlled
Brief Title: Prophylactic Antiemetic Efficacy of Palonosetron Versus Ondansetron for Cesarean Sections Under Regional Anesthesia
Acronym: PONV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, TSA, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Palonosetron01
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: PONV
Keywords: PONV; Palonosetron; Ondansetron; Cesarean section
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Sodium Chloride; Ondansetron; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Placebo Comparator): Patients in placebo group will receive spinal anesthesia with bupivacaine and morphine and a slow intravenous injection of saline 0,9%.
  Interventions: Drug: Ondansetron; Drug: Palonosetron
- Ondansetron group (Experimental): Patients in placebo group will receive spinal anesthesia with bupivacaine and morphine and a slow intravenous injection of ondansetron after cord clamping.
  Interventions: Drug: Placebo; Drug: Palonosetron
- Palonosetron group (Experimental): Patients in placebo group will receive spinal anesthesia with bupivacaine and morphine and a slow intravenous injection of palonosetron after cord clamping.
  Interventions: Drug: Placebo; Drug: Ondansetron

INTERVENTIONS:
Drug: Placebo — Patients will receive regular spinal anesthesia
  Other Names: Saline
  Arms: Ondansetron group; Palonosetron group
Drug: Ondansetron — Patients will receive slow intravenous injection of ondansetron 4 mg after cord clamping
  Arms: Palonosetron group; Placebo group
Drug: Palonosetron — Patients will receive slow intravenous infection of palonosetron 75 mcg after cord clamping
  Arms: Ondansetron group; Placebo group

SUMMARY:
This study aims to compare the quality of perioperative antiemesis of palonosetron and ondansetron in patients undergoing cesarean section

DETAILED DESCRIPTION:
Perioperative nausea and vomiting (PONV) related to spinal block anesthesia are common events and unpleasant for pregnant women. Its incidence can reach 80% in high-risk patients, and remains high despite the emergence of new antiemetic drugs.

Episodes untreated can result in prolonged stay in post-anesthetic care unit (PACU) and rehospitalization which can result in significant increase in overall costs of health care.

The purpose of the prophylaxis of PONV is therefore decrease its incidence, the stress of the patient, improve the quality and safety of surgical procedure and reduce hospital costs.

Antagonists of the 5-hydroxytryptamine 3 subtype receptor have been widely used and effective against PONV due to its efficacy and a favorable side-effect profile. Palonosetron is a new and potent drug generation5 second-HT antagonist with improved profile that acts longer. Recent studies where it was compared to ondansetron and palonosetron in high-risk patients in head and neck surgery and laparoscopic surgery is disclosed palonosetron far superior to ondansetron especially 2-24 hours after surgery. But there are no studies on caesareans comparing the two drugs.

This prospective, randomized, double-blind, placebo controlled, was designed to evaluate the efficacy of palonosetron compared with ondansetron and placebo for the prevention of nausea and vomiting in patients undergoing cesarean delivery under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I or II
* Scheduled for cesarean section on Maternal and Child Hospital of Brasilia, Federal District, Brazil

Exclusion Criteria:

* patients who had received antiemetics, diabetic, allergic to any study drug, corticosteroid use, psychoactive drugs, patients with vomiting in the course of gastrointestinal disease, eclampsia, heart disease, smokers, any evidence of fetal distress, psychiatric disease or who refused to participate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with nausea and vomiting | Within the first 48 hours after surgery

SECONDARY OUTCOMES:
Nausea Scores on the Number Rating Scale | Within the first 48 hours after surgery
  Quantify nausea by Number Rating Scale (NRS, ranging from 0 to 10 cm, zero being found when the patient is no nausea and ten, with maximum or un bearable nausea
Nausea Scores on the Verbal Rating Scale | Within the first 48 hours after surgery
  Verbal Rating Scale (VRS), consisting of a list of phrases (no nausea, mild nausea, moderate nausea, intense nausea, maximum nausea)
Apgar Newborn | delivery
  The resulting Apgar score ranges from zero to 10, measured at first and fifth minute
Likert Scale | 48 hours after surgery
  Overall satisfaction with the nausea - vomiting experience in a Likert scale of four points (dissatisfied, neutral, satisfied and very satisfied)
Number of participants with adverse events as a measure of safety and tolerability | delivery
  Intraoperative hemodynamic stability analysis through the incidence of tachycardia, hypertension, bradycardia, hypotension and consumed vasopressors
Number of participants with adverse events as a measure of safety and tolerability | Within the first 48 hours after surgery
  Incidence of adverse effects such as nausea, vomiting, pruritus, urinary retention, drowsiness and consumed rescue antiemetics

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonca, MD, TSA, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Chattopadhyay S, Goswami S. Palonosetron Versus Ramosetron Prophylaxis for Control of Postoperative Nausea and Vomiting after Cesarean Delivery under Spinal Anesthesia. J Obstet Gynaecol India. 2015 Feb;65(1):28-33. doi: 10.1007/s13224-014-0612-6. Epub 2014 Oct 7. PMID 25737619